CLINICAL TRIAL: NCT00051753
Title: A Multicenter, Randomized, Comparative Study to Evaluate the Efficacy and Safety of Levofloxacin in the Treatment of Children Who Have Recurrent and/or Persistent Acute Otitis Media
Brief Title: Levofloxacin In The Treatment Of Children With Recurrent And/or Persistent Acute Otitis Media
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004168
Record Dates: First submitted 2003-01-16; First posted 2003-01-17 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2011-01

CONDITIONS: Otitis Media
Keywords: Otitis Media; Acute Otitis Media; ear infection; levofloxacin; amoxicillin; clavulanate
MeSH Terms: conditions — Otitis Media; Otitis | interventions — Levofloxacin; Amoxicillin; Clavulanic Acid

INTERVENTIONS:
Drug: levofloxacin; amoxicillin/clavulanate

SUMMARY:
The purpose of this study is to demonstrate non-inferiority of levofloxacin compared with amoxicillin/clavulanate on the clinical response at the end of therapy in infants and children who have recurrent and/or persistent acute otitis media.

DETAILED DESCRIPTION:
This is a randomized, active-comparator, multicenter study consisting of 3 phases: a Pretreatment (Screening) Phase, a Treatment Phase, and a Posttreatment Phase. Subject eligibility will be determined at the screening visit based on signs and symptoms of acute otitis media (e.g., middle ear effusion, acute inflammation, acute purulent otorrhea) and criteria for recurrent and/or persistent acute otitis media. Eligible subjects will be randomized and drug will be dispensed by a study coordinator who will instruct parents and the subject about the importance of not revealing the assigned therapy to the subject's evaluator. Each subject will have an evaluator who will remain blinded to the subject's therapy throughout the study. Clinical assessments performed by a blinded evaluator at several time points throughout the study will be used to evaluate efficacy. Safety will be evaluated throughout the study by assessment of adverse events and changes in physical examinations (including musculoskeletal examination with evaluation of joints), vital signs, and clinical laboratory findings. Supplementary safety evaluations for musculoskeletal adverse events will be performed throughout the study. All subjects who enroll in this study and take at least 1 dose of levofloxacin or amoxicillin/clavulanate will be eligible to rollover into a long-term surveillance study primarily focused on the musculoskeletal system. The purpose of this study is to demonstrate non-inferiority of levofloxacin compared with amoxicillin/clavulanate on the clinical response at the end of therapy in infants and children who have recurrent and/or persistent acute otitis media. Either levofloxacin 10 mg/kg twice daily for 10 days (maximum daily dose of 500 mg) or amoxicillin/clavulanate (14:1) 45 mg amoxicillin/kg twice daily for 10 days (maximum daily dose of 3600 mg amoxicillin). Both study drugs will be given orally as a liquid suspension formulation

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged > or equal to 6 months to < 5 years
* Clinical signs and symptoms of otitis media including middle ear effusion and acute inflammation or acute purulent otorrhea
* At risk for difficult to treat Acute Otitis Media (AOM) is defined as having one of the following: recurrent Otitis Media (OM) as defined by 3 or more episodes in last 6 months or 4 or more episodes in past year or persistent OM as defined by evidence of AOM on 3rd day after starting any antimicrobial regimen
* Written consent/assent
* Have not participated in an experimental drug or medical device trial within 30 days prior to start of study.

Exclusion Criteria:

* History of hypersensitivity or serious reaction to any quinolone
* Tympanostomy tube in the affected ear
* Requires use of systemic antibiotic other than study drug
* Has a serious bacterial infection in addition to AOM that may interfere with assessment of their clinical response
* Diagnosed with bacterial meningitis
* Abnormal renal function defined as serum creatinine >0.5 mg/dL in infants 6 months or older and 0.8 mg/dL in children between 1 and 5 years of age
* History or presence of arthropathy or periarticular disease or any other musculoskeletal signs or symptoms that may confound a future safety exam of MS events
* Has a high probability of death during the study
* Poorly controlled seizure disorder or at risk for seizures
* HIV infection requiring pneumocystis carinii pneumonia prophylaxis
* Chronic use of corticosteroids 2mg/kg or more or 20mg/day for 14 or more days
* Amoxicillin/clavulanate (90 mg/kg/day) use within 3 days before the first dose of the study drug
* Previous participation in this protocol or another levofloxacin clinical study
* Employees of the investigator or study center with direct involvement in the study
* Family members are also excluded

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1643 (Actual)
Dates: Start 2002-11; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Clinical response (cured versus not cured) at Visit 3 (2 to 5 days after last dose).

SECONDARY OUTCOMES:
Clinical success (cured and improved versus failed) rate at Visit 3 (2 to 5 days after the last dose) and Visit 4 (10 to 17 days after the last dose); clinical cure rate at Visit 4 (10 to 17 days after the last dose); safety evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.